CLINICAL TRIAL: NCT06977022
Title: Clinical Trial on the Efficacy and Safety of Biodegradable 3D-Printed Implants in Chest Wall Reconstruction Surgery: A Prospective, Single-Arm Phase Il Study
Brief Title: Clinical Trial on the Efficacy and Safety of Biodegradable 3D-Printed Implants in Chest Wall Reconstruction Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202504-13
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chest Wall Tumor
Keywords: PCL Implant; Chest Wall Reconstruction; 3D Printing Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chest wall reconstruction (Experimental): Participants underwent extended resection of chest wall tumors followed by chest wall reconstruction using biodegradable polycaprolactone (PCL) 3D-printed rib implants.
  Interventions: Device: Chest wall reconstruction

INTERVENTIONS:
Device: Chest wall reconstruction — Extended resection of chest wall tumors with subsequent biodegradable polycaprolactone (PCL) 3D-printed rib prosthetic reconstruction

SUMMARY:
This project focuses on patients with chest wall tumors who are expected to have a maximum intraoperative anterolateral chest wall defect diameter of 5-10 cm and require chest wall reconstruction with rib implants. It aims to evaluate the efficacy and safety of biodegradable 3D-printed implants in chest wall reconstruction surgery, providing a superior reconstruction strategy for patients with tumor-induced chest wall defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria are eligible to participate in the study:

  1. Aged 18-70 years;
  2. No gender restriction;
  3. ECOG Performance Status 0-1;
  4. Chest CT-confirmed chest wall-originating tumor;
  5. Histologically/cytologically confirmed primary or metastatic chest wall tumor;
  6. Anticipated intraoperative anterolateral chest wall defect diameter 5-10 cm (maximum) or costal arch reconstruction required (investigator-assessed);
  7. Scheduled for prosthetic chest wall reconstruction;
  8. No prior chest wall reconstruction surgery;
  9. Willing to provide written informed consent and comply with follow-up visits and protocol requirements.

Exclusion Criteria:

* Patients who meet any of the following criteria are ineligible for this study:

  1. Patients with posterior chest wall defects;
  2. Uncontrolled underlying medical conditions or contraindications to general anesthesia;
  3. Pregnant or lactating women;
  4. Concurrent severe comorbidities that may interfere with study evaluations, including: Severe hepatic, cardiac, or renal diseases; Active malignancies (other than the indicated chest wall tumor); Alcohol use disorder
  5. lnability to provide reliable symptom reporting due to:P sychiatric disorders, Severe neurosis, Non-compliance with trial requirements
  6. Women of childbearing potential* and their partners unwilling to use effective contraception;
  7. Prior history of chest wall reconstruction surgery;
  8. Active uncontrolled bacterial, fungal, or viral infections;
  9. Participation in other clinical trials within 3 months prior to enrollment;
  10. Any other conditions deemedunsuitable by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Abnormal breathing | Postoperative 1 month, 3 months, 6 months, and 12 months
  Observe the integrity of the chest wall shape and the presence of abnormal breathing
Implant Degradation Performance Monitoring | Postoperative 1 month, 3 months, 6 months, and 12 months
  Thin-section chest CT + 3D imaging (DICOM format data)
  * Implant volume changes: Precise measurement of volumetric changes through 3D reconstruction;
    * Implant density changes: Quantification of density changes using Hounsfield Units (HU values), including adjacent bone tissue changes; ③ Bone resorption/formation: Observation of potential bone loss or new bone formation; ④ Implant structural integrity: Assessment for cracks, voids, or other structural compromises.
Peri-implant Soft Tissue Evaluation | Postoperative 1 month, 3 months, 6 months, and 12 months
  Chest MRI to evaluate thickening of the pleural fibrous layer surrounding the implant

SECONDARY OUTCOMES:
Changes in respiratory function--Pulmonary Function Test | Postoperative 1 month, 3 months, 6 months, and 12 months
  The assessment of changes in respiratory function through pulmonary function tests includes indicators such as Forced Vital Capacity (FVC), Forced Expiratory Volume in the First Second (FEV₁), Total Lung Capacity (TLC), Residual Volume (RV), and Maximum Voluntary Ventilation (MVV).
Adverse events | form date of enrollment until the end of the study, assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospitial, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No